CLINICAL TRIAL: NCT03340402
Title: Pilot Study of Preoperative Accelerated Partial Breast Irradiation for Triple Negative Breast Cancer Using Proton Beam Scanning
Brief Title: Preoperative Accelerated Partial Breast Irradiation for Triple Negative Breast Cancer Using Proton Beam Scanning
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Federal Share Core (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rachel Beth Jimenez, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-416; 208901 (Other: Federal Share Core); 2U19CA021239 (NIH)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Accelerated Partial Breast Irradiation (Experimental): Accelerated partial breast irradiation using proton beam scanning will consist of;
  * 5 daily treatments using custom prone patient immobilization, contrast-enhanced CT planning, and daily image guidance
  * Radiation therapy may be delivered with photons if proton treatments cannot be delivered
  * Dose will be prescribed such that the gross tumor (GTV) receives the prescription dose per institutional policy and standard of care
  * Daily target localization will also be confirmed using AlignRTTM
  Interventions: Radiation: Accelerated Partial Breast Irradiation; Device: AlignRT

INTERVENTIONS:
Radiation: Accelerated Partial Breast Irradiation — Proton radiation
Device: AlignRT — AlignRTTM uses infrared imaging to capture the 3D data of the patient's position to ensure accuracy of treatment delivery

SUMMARY:
This research study is studying an intervention as a possible treatment for Triple Negative Breast Cancer.

DETAILED DESCRIPTION:
This research study is a Pilot Study, which means this is the first time investigators are examining this study intervention in participants with triple negative breast cancer.

The FDA (the U.S. Food and Drug Administration) has not approved proton radiation for your specific disease but it has been approved for other uses.

The investigators believe that proton radiation administered in higher doses over a shorter time period may help stop cancer from growing while protecting the normal tissue cells.

In this research study, the investigators are researching how well proton radiation works in treating this type of breast cancer. Proton radiation is currently used in other types of breast cancer and the investigators believe that the higher doses of proton radiation administered over a shorter time period may lead to maximum efficacy in treating this type of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 40 years
* Core biopsy proven estrogen negative (< 1%), progesterone negative (< 1%), and HER2-neu negative (+1 by immunohistochemistry and/or FISH ratio < 2.0) invasive breast cancer
* Unicentric AJCC 7th edition T1N0M0 tumor measuring no greater than 2.0 cm in longest dimension on initial imaging with either breast MRI and/or mammogram
* ECOG Performance status < 1
* No prior treatment for this diagnosis of cancer
* No prior radiation to the ipsilateral breast, a history of contralateral breast radiation is permitted
* No clinical or radiographic evidence of malignant regional adenopathy
* No contraindication to breast conserving surgery, sentinel lymph node biopsy, or radiation therapy
* Ability to understand and willingness to sign a written informed consent document.
* Pregnant females are excluded. Female subjects of childbearing potential must indicate to their physician that there is not a possibility of being pregnant at the time of enrollment or have a negative pregnancy test prior to initiation of radiation therapy

Exclusion Criteria:

* Multicentric breast cancer, defined as discontiguous tumors separated by at least 5 cm of uninvolved tissue or discontiguous tumors that are located within separate breast quadrants either clinical or mammographically.
* Multifocal breast cancer, defined as discontiguous discrete foci of invasive carcinoma, separated by uninvolved intervening tissue, but within an overall span of 5 cm, or within the same breast quadrant.
* Tumor > 2.0 cm, nodal involvement, or metastatic involvement
* Patients with either diffuse (>1 quadrant or > 5 cm) suspicious microcalcifications on mammogram or diffuse non-mass-like enhancement on MRI
* History of ipsilateral cosmetic or reconstructive breast surgery
* Patients with a pacemaker or defibrillator
* Any contraindication to MRI including but not limited to the presence of a pacemaker/defibrillator or other implanted ferromagnetic device or an inability to lie prone
* Pregnant or lactating women
* Medical condition including but not limited to ongoing or active infection or connective tissue disease (e.g. systemic sclerosis or other collagen vascular diseases) that would, in the opinion of the treating physician, make this protocol unreasonably hazardous to the patient.
* Psychiatric illness/social situation that would limit ability to provide informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of grade ≥ 3 acute dermatitis | 4 Months
  The number of participants that experience grade 3 or greater acute dermatitis as assessed by Common Terminology Criteria for Adverse Events (CTCAE v4).

SECONDARY OUTCOMES:
The margins needed around Gross Tumor Volume (GTV) | 4 Months
  Summary of the margins needed around gross tumor volume based on the true tumor location.
Summary of treatment related adverse events | 2 years
  Summary of the treatment related adverse events experienced by participants as assessed by Common Terminology Criteria for Adverse Events (CTCAE v4)
Pathological response rate | 2 years
  Evaluation of the extent of residual active tumor following radiation as assessed on the surgical pathology specimen
Rates of local failure | 2 years
  The number of participants with local recurrence of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B Jimenez, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No